CLINICAL TRIAL: NCT06285630
Title: The Development and Health of the Intestinal Flora During the First Year of Life
Acronym: PREVENT
Status: Enrolling by invitation | Type: Observational
Sponsor: Alba Health AB (Industry)
Collaborators: Universiteit Antwerpen (Other); Uppsala University (Other); Copenhagen Studies on Asthma in Childhood (Other)
Responsible Party: Sponsor
Other Study IDs: Alba101; 2023-05299-01 (Other: Ethix)
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Healthy; Microbial Colonization
Keywords: Microbiome, Infant, healthy
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health infants: We aim to recruit parents of infants in an age range between 3 and 12 months. Healthy infants only, which were delivered in term, and that are not undergoing any antibiotic treatment.
  Interventions: Other: Observational, no intervation will be made

INTERVENTIONS:
Other: Observational, no intervation will be made — No intervention will be made, only longitudinal sample collection.

SUMMARY:
In this research study (PREVENT 1), Alba Health, in collaboration with academic institutions (Uppsala University, COPSAC and University of Antwerp) is investigating the association between the developing gut microbiota (collection of microbes present in the human gut) in the first year of life and lifestyle, wellbeing and health in a Swedish population. The study is the first of its kind in a Swedish population to collect and associate microbiome composition to an extensive family history and health questionnaire, stool colour and crying type, building on learnings from previous studies performed in other countries, such as the HELMI and COPSAC studies (HELMI - Finnish Health and Early Life Microbiota cohort from the University of Helsinki in Finland; COPSAC - Copenhagen Prospective Studies on Asthma in Childhood in Denmark).

The PREVENT 1 study is an observational research study led by Alba Health involving 300 families in Sweden with children between 0 and 12 months of age at the time of the study's start. After providing informed consent, the participating families will be asked to provide three stool samples from their child (the sample collection is not invasive and does not cause discomfort) and will be asked to answer questionnaires on lifestyle, well-being and family health. The participating families will not be asked to change their lifestyle beyond sample and data collection.

From the collected stool samples, we will extract microbial DNA and subject this to deep metagenomic sequence analysis. The study will only analyze microbial DNA, any human related material will be discarded. The stool samples will be destroyed within one month of sequencing (maximum 3 months from collection). The data will be stored according to GDPR and Swedish law, with informed consent in Sweden and with appropriate security measures. All research will be carried out in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants, no preterm and not undergoing antibiotic treatment

Exclusion Criteria:

* Preterm delivered infants or infants undergoing antibiotic treatment

Ages: 3 Months to 12 Months | Sex: All
Age Groups: Child
Study Population: We aim to recruit parents of infants in an age range between 3 and 12 months. Healthy infants only, which were delivered in term and that are not undergoing any antibiotic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-26 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Microbiome composition of infants in variable age ranges | 3 times points with 3 months in between time points
  How the microbiome changes according to age

SECONDARY OUTCOMES:
Is the composition associated with and gastrointestinal issues | 3 times points with 3 months in between time points
  How the microbiome composition in different ages can be associated with different GIT disturbances in infants between 3 and 12 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Willem M de Vos, PhD, Principal Investigator — Alba Health AB
Locations (1):
- Alba Health AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
We will make the metagenomic sequences publicly available upon publication as required by all scientific journals but no other IPD will be published in line with the GDPR requirements